CLINICAL TRIAL: NCT03425864
Title: Pink Esthetic Score Evaluation After Soft Tissue Augmentation Using Connective Tissue Graft Around Immediate Dental Implants Versus Immediate Dental Implants Alone in Esthetic Zone
Brief Title: PES After Soft Tissue Augmentation Using CTG Around Immediate Dental Implants Versus Immediate Dental Implants Alone in Esthetic Zone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nada Farouk Hasan Abd El-Aziz (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, Nada Farouk Hasan Abd El-Aziz, Assistant Specialist, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2010
Record Dates: First submitted 2018-01-26; First posted 2018-02-08 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2020-10

CONDITIONS: Soft Tissue Augmentation
Keywords: immediate implant; connective tissue graft
MeSH Terms: interventions — Immediate Dental Implant Loading

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomized using sequence generation program (Random.org in equal proportions between control group (immediate implant alone) and study group (immediate implant covered with sub-epithelial connective tissue graft with full coverage technique).
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blinded Blinding will be done to the clinical, radiographic assessors, without involving them in sequence generation or allocation concealment or surgery performing.
  Blinding of the biostatistian.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- immediate implant (Other): patient will receive immediate implant alone.
  Interventions: Device: immediate implant
- immediate implant with connective tissue graft (Active Comparator): patient will receive immediate implant and connective tissue gaft
  Interventions: Procedure: connective tissue graft; Device: immediate implant

INTERVENTIONS:
Procedure: connective tissue graft — patient will receive immediate implant and connective tissue graft
  Other Names: subepithelial connective tissue graft
  Arms: immediate implant with connective tissue graft
Device: immediate implant — patient will receive immediate implant with connective tissue graft.
  Other Names: post extraction dental implant

SUMMARY:
The goal of the present study is to compare the esthetic result and stability of gingival tissue over the immediate implant only and immediate implant with connective tissue in patients with single non-restorable tooth in the esthetic zone. The main null hypothesis to be tested is that the addition of SCTG to immediately placed implants will not significantly differ from immediately placed implant alone as regard gingival tissue stability.

DETAILED DESCRIPTION:
Implant became a treatment modality for replacing missing or non-restorable teeth, providing clinical success rate and esthetic outcome. (1) In esthetic zone the main goal is not only the preservation of function but also the preservation of the esthetics. The esthetic outcome of implant supported restoration depend on the soft tissue volume and the soft tissue contour. (2) The placement of immediate implant after tooth extraction was proved as a very high success rate treatment modality. It provided several advantages such as reduction of the time between tooth extraction and the placement of prosthesis, reduction of the number of surgical treatments (3) and increase osteointegration between bone and implant surface (4).

Considering the survival rate of immediate implantation versus delayed implantation there is no significant difference with an overall success rate of 99.6%, it is just considered as a successful treatment modality, based on 802 implants (5).

On the other hand disadvantage related to esthetic outcome has been reported, showing facial gingival recession following the first year of function due to labial bone plate resorption. (6, 2).

A systematic review by Sanz et al.,(2012) compared the reduction of bone height and bone width between two groups the control group was delayed implant placement and the studied group was immediate implant placement and the mean difference between groups was of 13.11% (95% CI: from 3.83 to 22.4; P = 0.057) and 19.85% (95% CI: from 13.85 to 25.81)respectively, concluding that the early placement of dental implants after tooth extraction offers advantages in terms of soft and hard tissue preservation, compared with delayed implant placement , which affect the aesthetic (7 ) As a sequence of dimensional ridge alterations that occur following tooth extraction many studies reported a recession of marginal peri-implant mucosa, which affect the aesthetic outcome (8, 9, and 10).

A study made by Migliorati et al., (2015) between two groups, the control group (immediate loading implant treated without raising a flap) and the test group (immediate loaded implant treated with sub-epithelial connective tissue graft (SCTG) using the tunnel technique in the labial area) Both groups (47 implants) received deproteinized bovine bone minerals and implants were successfully integrated with a follow up period 2-year examination . Moreover the mean recession in the control group was 0.71mm (17.58%), one third of the control group reported recession >1mm, and mean pink aesthetic score (PES) was 6.65, resulting in bad aesthetic. The test group showed an increase of the keratinized mucosa (KM) with a mean of 34.29% (0.5mm) and a mean recession of 0.2mm (10.01%), only one case (4%) showed recession >1mm and the mean PES was 8. The thickening of soft tissue by the addition of SCTG, lead to compensation and maintenance of the loss of bone volume in the labial area (11).

The addition of sub epithelial connective tissue graft (SCTG) to the immediate implant was suggested for facial gingival biotype conversation. It was proved to be successful in preserving soft tissue levels. (12)

A systematic review was made to investigate if the addition of SCTG overcome the disadvantage of placement of immediate implant only or not, but unfortunately the included studies had different techniques and the number of the patients in those studies was few thus further RCT was necessary (13).

ELIGIBILITY:
Inclusion Criteria:

Non-restorable teeth located within the maxillary anterior area and premolars. Age ranged between 20 to 50 years old. Sufficient vertical inter-arch space upon centric occlusion. Patients with good oral hygiene. Intact labial/buccal bone plate.

10. a. Inclusion criteria

1. Age: 20-50. 2. Patients with single non-restorable teeth in anterior or premolar area. 3. "Patients with adequate bone volume for the dental implant procedure". 5. Patients who are compliant to oral hygiene measures. 6. Patient consent approval and signing.

10. b. Exclusion criteria:

1. Patients with any systemic disease that could affect normal healing of tissue and predictable outcome.
2. Patients with any habits that might affect osseointegration, such as heavy smoking and alcoholism.
3. Pregnant women.
4. Patients with untreated periodontal disease or the presence of pathologic condition at implant site.
5. Patients with Parafunctional habits that produce overload on the implant such as bruxism and clenching.
6. Shallow palate.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2020-09-13 (Actual); Study Completion 2020-10-13 (Actual)

PRIMARY OUTCOMES:
pink esthetic score | should be measured after 8 months below implant and graft placement
  evaluation of pink esthetic score around immediate implant only in esthetic zone around immediate implant with connective tissue graft in esthetic zone

SECONDARY OUTCOMES:
tissue piotype | should be measured after 6 months below implant and graft placement
  It is measured by penetrating the gingiva perpendicular to the tooth with the periodontal probe down to the bone after giving local anesthesia to determine the thickness of the tissue and apical to the gingival margin at the vertical bisecting midline with reference to the cementoenamel junction of adjacent teeth.
width of keratinized gingiva | should be measured after 6 months below implant and graft placement
  It is recorded as the distance from the mucogingival junction (MGJ) to the free gingival margin of the related tooth by graduated periodontal probe.

CONTACTS AND LOCATIONS:
Locations (1):
- Nada Abd El Aziz, Minya, Minya Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No